CLINICAL TRIAL: NCT01593683
Title: Waitlist-controlled Trial of a Psychological Education Program for Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William Pirl, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MGH 2011-P-002799
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Psychological Stress
Keywords: Oncology service; Nursing staff; Psychosocial intervention; Coping skills
MeSH Terms: conditions — Stress, Psychological; Neoplasms | interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychological education program (Experimental): Patients receive the psychological education program upon study enrollment.
  Interventions: Behavioral: Psychological education program for nurses
- Waitlist (No Intervention): Participants are assigned to a 16-week wait-list period upon enrollment. Participants are invited to receive the psychological education program following the waitlist period.

INTERVENTIONS:
Behavioral: Psychological education program for nurses — Approximately 4 weekly one-hour group sessions led by study clinicians and 1 optional individual session with a single study clinician.
  Arms: Psychological education program

SUMMARY:
The purpose of this study is to test a brief education program for oncology nurses, to enhance their skills for managing psychosocial stressors associated with providing direct patient care. The investigators will explore efficacy of the intervention for reducing psychological stress and medical errors.

ELIGIBILITY:
Inclusion Criteria:

* Must have RN degree
* Must be employed as an oncology nurse in an inpatient, infusion, or ambulatory care unit

Exclusion Criteria:

* Participation in earlier pilot trial of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in psychological stress as measured by the Perceived Stress Scale and the Maslach Burnout Inventory | At approximately 16 and 32 weeks post-baseline

SECONDARY OUTCOMES:
Change in from baseline in medical errors as measured by the Medical Errors Questionnaire | At approximately 16 and 32 weeks post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: William F Pirl, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States